CLINICAL TRIAL: NCT05687825
Title: Operative Risk Factors for Clinically Relevant Postoperative Pancreatic Fistula After Pancreaticoduodenectomy: A Prospective Multicenter Cohort Study
Brief Title: Risk Factors for Clinically Relevant Postoperative Pancreatic Fistula
Status: Completed | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, MD, Associate professor of surgery, South Valley University
Other Study IDs: SVU/MED/SUR011/4/23/4/612
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Fistula
Keywords: risk factors,; clinically relevant pancreatic fistula,; pancreaticoduodenectomy
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinically relevant postoperative pancreatic fistula: patients who developed clinically relevant postoperative pancreatic fistula after pancreaticoduodenectomy
  Interventions: Procedure: pancreaticoduodenectomy procedure
- No clinically relevant postoperative pancreatic fistula: patients who did not develop clinically relevant postoperative pancreatic fistula after pancreaticoduodenectomy
  Interventions: Procedure: pancreaticoduodenectomy procedure

INTERVENTIONS:
Procedure: pancreaticoduodenectomy procedure — Pancreaticoduodenectomy operation

SUMMARY:
For periampullary and pancreatic head disorders, pancreaticoduodenectomy (PD) is the standard treatment. However, PD is technically demanding and has high morbidity and mortality rates. The most significant and life-threatening complication of PD is postoperative pancreatic fistula (POPF), with reported rates of 5 to 70% for total POPF and 10 to 45% for clinically relevant (CR-POPF). Operative risk variables for CR-POPF after PD were investigated in this study.

DETAILED DESCRIPTION:
For periampullary and pancreatic head disorders, pancreaticoduodenectomy (PD) is the standard treatment. However, PD is technically demanding and has high morbidity and mortality rates. The most significant and life-threatening complication of PD is postoperative pancreatic fistula (POPF), with reported rates of 5 to 70% for total POPF and 10 to 45% for clinically relevant (CR-POPF). Operative risk variables for CR-POPF after PD were investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with resectable distal CBD carcinoma, periampullary carcinoma, duodenal carcinoma, and carcinoma of the head of the pancreas.
2. American Society of Anesthesiologists (ASA) scores I & II.
3. Patients aged > 20 years.
4. Agreement to complete the study.

Exclusion Criteria:

1. Patients with benign disease, trauma, and receive neoadjuvant therapy.
2. double primary cancers.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — more than 20 years
Study Population: all consecutive patients who were treated with a pancreaticoduodenectomy
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
clinically relevant post operative pancreatic fistula | 10 days
  A drainage fluid of any measurable volume with an amylase level more than three times the upper normal serum level on or after the 3rd postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Omar, M.D., Principal Investigator — General Surgery Department, Faculty of Medicine, South Valley University
Locations (1):
- Qena faculty of Medicine, South Valley University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No